CLINICAL TRIAL: NCT03599531
Title: A Pilot Study to Evaluate the Utility of the SomaLogic Cardiovascular Disease (CVD) Secondary Risk Panel as a a Tool to Stratify Cardiovascular Risk
Brief Title: Utility of the SomaLogic Cardiovascular Disease (CVD) Secondary Risk Panel for Cardiovascular Risk
Status: Completed | Type: Observational
Sponsor: SomaLogic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLI1002F011
Record Dates: First submitted 2018-05-25; First posted 2018-07-26 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Risk Factor; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA plasma blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective pilot study of participants who have stable coronary heart disease (CHD). Participants undergo risk stratification using the SomaLogic Cardiovascular Disease (CVD) Risk Panel blood test at baseline and again 4-12 months after the initial test. Participant surveys and chart abstractions are conducted at baseline and follow-up to collect feedback about the test report and actions taken. Care teams may consider using the risk information from the SomaLogic panel to address care gaps. Medical treatment decisions and recommendations are confirmed by established clinical methods, including blood pressure monitoring, body mass index (BMI), lipid and c-reactive protein (CRP) measurements, and physician's clinical judgment.

DETAILED DESCRIPTION:
This is a prospective pilot study of participants who have stable coronary heart disease (CHD). Objectives of this study are to understand whether CVD Secondary Risk Panel scores change from baseline to follow-up (4-12 months after baseline) and actions taken, if any, based upon the results. Participants are surveyed to learn what the test results mean to them and assess if the results affect adherence to therapy and lifestyle choices (diet, exercise, alcohol, and tobacco use). In addition, this study will investigate the characteristics of patients that physicians choose to test with the CVD Secondary Risk Panel, and what actions the care team takes because of the results of the test. Medical treatment decisions and recommendations are confirmed by established clinical methods, including blood pressure monitoring, BMI, lipid and CRP measurements, and physician's clinical judgement. Chart abstractions and participants surveys occur at the baseline and follow-up visits, and charts may be abstracted annually for up to 10 years post enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 40
* Stable CHD documented by at least one of the following: history of myocardial infarction >6 months prior to study enrollment, angiographic evidence of at least 50% stenosis, abnormal CAC score, prior evidence of inducible ischemia by treadmill or nuclear testing, or a history of coronary revascularization
* Ability to provide informed consent

Exclusion Criteria:

* Inability or unwillingness to provide informed consent
* Less than 40 years of age
* History of myocardial infarction in the prior 6 months.
* Treatment for malignancy (other than basal or squamous cell carcinomas of the skin) within the last 2 years
* Pregnancy
* Individuals deemed ineligible by the Investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be 40 years or older with stable Coronary Heart Disease (CHD)
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Decrease in SomaLogic CVD Secondary Risk Score from baseline to follow-up. | 12 months
  Percent of participants whose CVD risk score decreased from baseline to follow-up. This is assessed on a numeric scale of 1 (lower risk) to 5 (higher risk).

SECONDARY OUTCOMES:
Motivation for adherence to medication assessed by a self-reported questionnaire. | 12 months
  Impact of the CVD Secondary Risk Score on patient adherence to therapy. Assessed by percent of patients whose motivation to adhere increased on a 5-point scale from baseline to follow-up.
Motivation for a healthy diet assessed by a self-reported questionnaire. | 12 months
  Impact of the CVD Secondary Risk Score on diet. Assessed by percent of patients whose motivation for a healthy diet increased on a 5-point scale from baseline to follow-up.
Motivation for exercise assessed by a self-reported questionnaire. | 12 months
  Impact of the CVD Secondary Risk Score on exercise. Assessed by percent of patients whose motivation to exercise increased on a 5-point scale from baseline to follow-up.
Motivation for decreased alcohol use assessed by a self-reported questionnaire. | 12 months
  Impact of the CVD Secondary Risk Score on alcohol use. Assessed by percent of patients whose alcohol use decreased on a 5-point scale from baseline to follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Williams, MD, PhD, Principal Investigator — SomaLogic, Inc.
Locations (1):
- Boulder Heart, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No